CLINICAL TRIAL: NCT05875922
Title: Prospective Post-Market Clinical Follow-Up (PMCF) Study to Investigate the Clinical Outcomes of a ISOPURE and EYHANCE Intraocular Lenses (IOL)
Brief Title: Comparison of ISOPURE and EYHANCE (Switzerland)
Acronym: PHY2301
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHY2301
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular Lens; EDOF; hydrophobic; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind masking; Patient will not be informed which IOL model was implanted until end of the study. Outcomes assessors will not be informed which IOL model was implanted until end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): Experimental arm: Premium monofocal intraocular lens.
  Interventions: Device: IOL implantation experimental (ISOPURE 1.2.3.)
- IOL implantation active comparator (Active Comparator): Comparator arm: EDOF intraocular lens.
  Interventions: Device: IOL implantation active comparator (TECNIS Eyhance)

INTERVENTIONS:
Device: IOL implantation experimental (ISOPURE 1.2.3.) — Implantation of premium monofocal IOL ISOPURE 1.2.3.
  Arms: IOL implantation experimental
Device: IOL implantation active comparator (TECNIS Eyhance) — Implantation of EDOF IOL TECNIS Eyhance
  Arms: IOL implantation active comparator

SUMMARY:
This is a prospective randomised open-label study with the aim to compare the visual performance of the premium monofocal Isopure IOL versus the extended depth of focus Eyhance® IOL after phaco-emulsification cataract surgery.

DETAILED DESCRIPTION:
This is a single center, prospective, randomised, controlled, double-blind post-market clinical follow-up (PMCF) study whereby patients undergoing routine cataract surgery will have bilateral implantation of premium monofocal intraocular lenses (PhysIOL ISOPURE 1.2.3.) or EDOF lenses (TECNIS Eyhance). The patients will be randomized in a 1:1 ratio to receive the study or control lenses. Both IOLs, investigational device and control device, are CE approved and commercially available in the countries this clinical investigation is being carried out. The investigational device and all study products, including the devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

The device under investigation (ISOPURE 1.2.3.) is a hydrophobic, glistening-free, acrylic premium monofocal intraocular lens (IOL) manufactured by the sponsor of this study, PhysIOL sa/nv. The control lens (TECNIS Eyhance) is a non-diffractive Extended Vision Posterior Chamber IOL.

The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

Subjects participating in the trial will attend a total of 6 study visits (1 preoperative, 1 operative and 4 postoperative) over a period of 6 months. Subjects would have the option for unscheduled visits if required medically.

Primary and secondary endpoint data will be collected at the 120-180 days follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity;
* Calculated IOL power is within the range of the study IOLs;
* Male or female adults ages 50 years or older on the day of screening who have cataract(s) in one or both eyes;
* Regular total corneal astigmatism ≤1.0 D (measured by topography method)
* Clear intraocular media other than cataract;
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures;
* Expected postoperative Best Corrected Distance Visual Acuity (CDVA) ≤ 0.2 logMAR;
* Signed informed consent.

Exclusion Criteria:

* Age of patient < 50 years;
* Regular total corneal astigmatism >1.0 dioptres (measured by topography method)
* Irregular astigmatism;
* Difficulty for cooperation (distance from their home, general health conditions);
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders);
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema or macula pucker; previous laser treatment for peripheral retinal tears is allowed;
* Previous intraocular or corneal surgery or intravitreal injection;
* Traumatic cataract;
* History or presence of macular edema;
* Glaucoma with visual field defects; or RNFL defects on OCT; ocular hypertension is allowed;
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic / scotopic conditions);
* Amblyopia with monocular preoperative CDVA of >0.1 logMAR;
* Cornea guttata;
* Keratoconus;
* Chronic uveitis;
* Expected complicated surgery;
* Significant dry eye;
* Contra-indications as listed in the current Instructions for use (IFU);
* Contra-indication or unwillingness to perform immediate sequential bilateral cataract surgery;
* Concurrent or previous (within 60 days) participation in another drug or device investigation.

In addition to above mentioned in- and exclusion criteria, subjects shall be discontinued when certain conditions are present at the time of surgery, including:

* zonular instability or defect;
* capsular fibrosis or other opacity; and
* inability to fixate IOL in desired position. In such cases, the subject shall be followed until the condition has stabilized.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
monocular Best Corrected Distance Visual Acuity (CDVA) under photopic light conditions on the first implanted eye. | 6 months (120-180 days) postoperative
  Non inferiority of ISOPURE 1.2.3. outcomes compared to the TECNIS Eyehance outcomes in terms of monocular Best Corrected Distance Visual Acuity (CDVA) by means of statistical significance.
  A significance level of 0.05 or lower (p < 0.05) will be considered statistically significant. CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018.

SECONDARY OUTCOMES:
Safety (Rates of Adverse Events) | 1 day (1-2 days) postoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The objective is to compare the SPE (Safety and Performance Endpoints) rates of the investigational product to the results of historical data of EN ISO 11979-7:2018, Annex E (Table E.2)

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Preoperative, 1 day (1-2 days) postoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Anterior Chamber Depth | Preoperative
  Anterior Chamber Depth measurement is performed using the IOLMaster device. This measurement is required to calculate the required IOL power. The measurement unit is mm. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Axial Lenght | Preoperative
  Axial Length measurement is performed using the IOLMaster device. This measurement is required to calculate the required IOL power. The measurement unit is mm. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Lens Thickness | Preoperative
  Lens Thickness measurement is performed using the IOLMaster device to asses the dimension of the natural lnes. This measurement is required to calculate the required IOL power. The measurement unit is mm. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry measurement - K values | Preoperative
  Keratometric measurements are performed to calculate the required IOL power. The measurement is performed using the IOLMaster device. This specific outcome measure is to measure the K value in the steep axis (K1) and flat axis (K2). The measurement unit is diopter (D). The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power | Operative (day of surgery)
  The IOL spherical power of the implanted IOL must be recorded.
Target refraction | Operative (day of surgery)
  The target refraction given by the IOL calculator must be recorded. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Preoperative, 1 month (30-60 days) postoperative
  An OCT (optical coherence tomography) image will be taken at the preoperative visit and 1 months postoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size under mesopic light conditions | preoperative
  Mesopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Manifested refraction | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | Preoperative, 1 day (1-2 days) postoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  monocular and binocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Binocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) under mesopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Binocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done binocularly under mesopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 6 months (120-180 days) postoperative
  Binocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA@66cm) under photopic light conditions | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular DCIVA@66cm is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity at 66cm (UIVA@66cm) under mesopic light condition | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Binocular UIVA@66cm is measured with ETDRS charts placed in 66cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done binocularly under mesopic light conditions.
Monocular Distance Corrected Near Visual Acuity at 40cm (DCNVA) under photopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Near Visual Acuity at 40cm (UNVA) under photopic light conditions | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular UNVA is measured with ETDRS charts placed in 40cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Binocular Defocus Curve | 1 month (30-60 days) postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -2.5 D to +1.5 D in 0.5 D steps. This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions | 6 months (120-180 days) postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device CSV-1000 (Vector Vision). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 6 months (120-180 days) postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (Vector Vision). This examination is performed binocularly.
Slitlamp examination - Corneal status | Preoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Slitlamp examination - Signs of inflammation | Preoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Signs of inflammation
Slitlamp examination - Iris status | Preoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Iris status
Fundus examination with dilated pupil | Preoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Optic nerve cupping | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Optic nerve cupping
Slitlamp examination - Posterior Capsular Opacification (PCO) or Posterior Capsular Fibrosis | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Posterior Capsular Opacification (PCO) or Posterior Capsular Fibrosis
Slitlamp examination - IOL discoloration | 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL discoloration.
Slitlamp examination - abnormal IOL positioning | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - abnormal IOL positioning
Patient reported outcomes - Quality of Vision questionnaire | 6 months (120-180 days) postoperative
  To assess the subjective perception of disturbances by photic phenomena. Subjects answer one question per category on their individual perception of glare, halo and starbursts, respectively. Answers are graded in 5 steps between always and never.
  Descriptive analysis will be performed on the occurence of photic phenomena per category. This questionnaire does not consist of a scaling.
Patient reported outcomes - Patient-Reported Spectacle Independence Questionnaire (PRSIQ) [Morlock et al, 2017] | 6 months (120-180 days) postoperative
  The Patient-Reported Spectacle Independence Questionnaire (PRSIQ) is a patient-reported measure assessing spectacle independence following cataract surgery. The analyses conducted provide evidence for the use of the PRSIQ total score as a measure of spectacle independence [Morlock et al, 2017].
  In the first category, subjects are asked if they need glasses for distance vision, intermediate vision and near vision with 'yes' and 'no' being the only possible answers.
  In the second category, patients are asked to scale their frequency of using spectacles over the last 7 days for three different distances with 5 ratings ranging from '1: All of the time' to '5: None of the time'. A higher rating means higher rate of spectacle independence.
  In addition, patients are asked to scale if they are able to function without spectacle aid for three different distances with 5 ratings ranging from '1: All of the time' to '5: None of the time'. A higher rating means higher rate of spectacle freedom.

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Vandekerkchove, MD, Principal Investigator — Eye center Vista Alpina
Locations (1):
- Eye center Vista Alpina, Visp, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605
- [Background] Tomagova N, Elahi S, Vandekerckhove K. Clinical Outcomes of a New Non-Diffractive Extended Depth-of-Focus Intraocular Lens Targeted for Mini-Monovision. Clin Ophthalmol. 2023 Mar 25;17:981-990. doi: 10.2147/OPTH.S405267. eCollection 2023. PMID 37007049
- [Background] Auffarth GU, Gerl M, Tsai L, Janakiraman DP, Jackson B, Alarcon A, Dick HB; Quantum Study Group. Clinical evaluation of a new monofocal IOL with enhanced intermediate function in patients with cataract. J Cataract Refract Surg. 2021 Feb 1;47(2):184-191. doi: 10.1097/j.jcrs.0000000000000399. PMID 32932369
- [Background] Wan KH, Au ACK, Kua WN, Ng ALK, Cheng GPM, Lam NM, Chow VWS. Enhanced Monofocal Versus Conventional Monofocal Intraocular Lens in Cataract Surgery: A Meta-analysis. J Refract Surg. 2022 Aug;38(8):538-546. doi: 10.3928/1081597X-20220707-01. Epub 2022 Aug 1. PMID 35947003